CLINICAL TRIAL: NCT03255447
Title: Phase II Trial Investigating the Safety and Feasibility of Peptide GAM Immunoadsorption in Anti-PLA2R Positive Autoimmune Membranous Nephropathy
Brief Title: Peptide GAM Immunoadsorption Therapy in Autoimmune Membranous Nephropathy
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Fresenius AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R04240
Record Dates: First submitted 2017-08-11; First posted 2017-08-21 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Autoimmune Membranous Nephropathy
Keywords: Idiopathic Membranous Nephropathy; Primary Membranous Nephropathy; Immunoadsorption; Apharesis
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunoadsorption therapy (Experimental): Peptide GAM immunoadsorption therapy
  Interventions: Device: Immunoadsorption

INTERVENTIONS:
Device: Immunoadsorption — Fresenius Globaffin

SUMMARY:
Autoimmune Membranous Nephropathy is now understood to be a condition caused by the immune system although the exact mechanism is not completely known. This study aims to remove the offending part of the immune system using immunoadsorption to not only treat the disease but also use the opportunity to better understand the mechanism of disease. This will allow more targeted treatment in the future with less complications and side effects.

DETAILED DESCRIPTION:
Membranous nephropathy (MN) is among the most common causes of nephrotic syndrome in adults worldwide. The majority of patients will remain stable with either complete remission or partial remission but approximately 20% will progress slowly to end stage renal disease necessitating the need for renal replacement therapy (RRT).

Current standard therapy for primary (or autoimmune) membranous nephropathy is a regime of rotating high dose steroids and immunosuppression was first described in the mid-nineties and has been the mainstay of treatment since but comes with a high side effect burden.

Idiopathic membranous nephropathy is now understood to be an autoimmune disease characterised by the presence of IgG autoantibodies to M-Type Phospholipase A2 Receptor (anti-PLA2R). Immunoadsorption is a method of removing specific circulating immunoglobulins and has been shown to remove over 80% of circulating IgG with a single session immunoadsorption of 2.5 plasma volumes, with albumin and antithrombin III almost unaffected. With multiple sessions this can rise to over 98%.

Immunoadsorption therapy has been in use for a number of years and this study will use Peptide GAM Immunoadsorption therapy developed by Fresenius Healthcare. This uses two systems, the Art Universal and ADAsorb. The Art Universal became commercially available in 2005 and the ADAsorb in 2002.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed Primary Membranous Nephropathy within the last 3 years
* Active disease despite 6 months of supportive care including ACEi or ARB (Active disease defined as uPCR > 300mg/mmol or 24 hour urinary protein >3.5g/1.73m2)
* Disease severity that in the physicians view warrants treatment prior to completion of 6 months supportive care
* Anti-PLA2R titre > 170 u/ml
* Haemophilus and Pneumococcal vaccinations up to date
* Above the age of 18
* Able to provide informed consent

Exclusion Criteria:

* Evidence of causes of secondary membranous nephropathy
* eGFR < 20ml/min
* Treatment with steroids or immunosuppression (including but not limited to cyclophosphamide, MMF or azathioprine) and Biologics (including but limited to Rituximab or belimumab) within 6 months of screening
* Therapeutic Plasma Exchange within 28 days of screening
* Previous renal transplantation
* Co-morbidity, which in physicians' view, would preclude patient from treatment with immunoadsorption.
* Pregnant at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Serum anti-PLA2R titres | 14 days
  Reduction in serum anti-PLA2R titres to normal range

SECONDARY OUTCOMES:
The incidence of treatment related adverse events as defined by CTCAE v4.0 | Day 14, 28, 56, 84, 168 and 365
  To assess the safety and tolerability of Immunoadosorption therapy
To determine the effect on disease activity (efficacy) | Day 14, 28, 56, 84, 168 and 365
  Assessment of reduction in proteinuria level and change in eGFR from baseline
Serum anti-PLA2R titres | Day 14, 28, 56, 84, 168 and 365
  Kinetic modelling of serum anti-PLA2R levels
To determine the effect on Quality of life measures (EQ5D) | Day 14, 28, 56, 84, 168 and 365
  To determine the effect on Quality of life measures (EQ5D)
Cost-effectiveness | Day 14, 28, 56, 84, 168 and 365
  Cost-effectiveness of treatment (Incremental cost-effectiveness ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Mitra, Principal Investigator — Central Manchester University Hospital Foundation Trust
Locations (3):
- United Kingdom (3):
  - Central Manchester University Hospital Foundation Trust, Manchester, Greater Manchester
  - Royal Preston Hospital, Preston, Lancashire
  - Salford Royal Infirmary, Salford, Lancashire

IPD SHARING:
Plan to Share IPD: No